CLINICAL TRIAL: NCT02919254
Title: Evaluation of Various Doses of Beetroot Juice on Anaerobic Performance
Brief Title: Beetroot Juice Doses and Anaerobic Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Semone Myrie, Dr. Semone Myrie, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: J2015:108
Record Dates: First submitted 2016-08-05; First posted 2016-09-29 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Anaerobic Exercise; Dietary Supplementations

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Dosage (Active Comparator): Subjects will receive approximately 8 mmol of dietary nitrate per day delivered as a commercially available beetroot juice supplement for 7 days.
  Interventions: Dietary Supplement: Beet It Sport Shot
- Moderate Dosage (Active Comparator): Subjects will receive approximately 0.5 mmol of dietary nitrate per day delivered as a commercially available beetroot juice supplement for 7 days.
  Interventions: Dietary Supplement: Beet It Sport Shot
- Placebo (Placebo Comparator): Subjects will receive a placebo beverage containing negligible nitrate for 7 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Beet It Sport Shot — Commercially available concentrated beetroot juice supplement intended for athletes.
  Arms: High Dosage; Moderate Dosage
Other: Placebo — Fruit juice cordial containing negligible nitrate
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effect of varying nitrate doses of beetroot juice supplementation on dynamic, multijoint resistance exercise performance in active, trained individuals. Performance will be assessed based on parameters including neuromuscular efficiency, anaerobic performance capability, oxygen consumption, plasma nitrate/nitrite levels, specific muscle tissue biomarkers including lactate, and anthropometric measurements of select muscle groups.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 6 consecutive months experience in resistance training, engaging at least 2 times per week.
* Possess sufficient mobility to properly execute movements required in testing protocol

Exclusion Criteria:

* Usage of any banned dietary supplements or performance enhancing drugs (thermogenics, anabolic steroids, prohormones, etc.)
* Any physical condition or malady that would impede participant from performing exercise or by doing so, endanger the individual

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2016-08; Primary Completion 2017-05 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Muscle activation and fiber recruitment | 5 weeks
  Muscle activation/fiber recruitment to be measured in millivolts (mV) using electromyography (EMG) sensor during maximum voluntary contractions (MVC) and compared between study arms.

SECONDARY OUTCOMES:
Plasma nitrate/nitrite levels | 5 weeks
  Plasma nitrate and nitrite levels will be measured at baseline and after 7 days of supplementation and compared between study arms.
Number of repetitions performed | 5 weeks
  Total number of repetitions in each session and number of repetitions performed at each respective % of 1 repetition maximum during each session will be recorded and compared between study arms.
Oxygen consumption | 5 weeks
  Total oxygen consumption during testing sessions will be recorded and compared between study arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No